CLINICAL TRIAL: NCT06343844
Title: Disparities in Myocardial Infarction Remodeling According to Gender
Acronym: REMOVE 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC23_0070
Record Dates: First submitted 2024-02-23; First posted 2024-04-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Myocardial Infarction; Ventricular Remodeling
Keywords: Non-Interventional Registry; Biorepository Establishment
MeSH Terms: conditions — Myocardial Infarction; Ventricular Remodeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- case control registry (Other): left ventricular remodeling measurement with cardiac echography
  Interventions: Diagnostic Test: cardiac imaging to assess left ventricular volumes and function

INTERVENTIONS:
Diagnostic Test: cardiac imaging to assess left ventricular volumes and function — non-invasive cardiac imaging (echocardiography and MRI)

SUMMARY:
Following myocardial infarction, female individuals demonstrate a poorer prognosis, characterized by elevated rates of mortality and heart failure. A primary hypothesis suggests unfavorable cardiac remodeling in women. This remodeling, defined as alterations in cardiac size and shape post-infarction, necessitates repeated non-invasive imaging for study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* First myocardial infarction with ST-segment elevation during the hospital phase
* Coronary angiography performed within 72 hours of the infarction
* Inclusion in the RIMA registry
* Patient affiliated or beneficiary of a social security scheme; Signature of informed consent

Exclusion Criteria:

* Patients already enrolled in the study
* Poor understanding of the French language
* Pregnant, breastfeeding, or postpartum women
* Individuals deprived of liberty by judicial or administrative decision; Individuals receiving psychiatric care under coercion
* Individuals subject to a legal protection measure; Individuals incapable of giving consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1650 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2039-11-01 (Estimated); Study Completion 2040-09-01 (Estimated)

PRIMARY OUTCOMES:
Asses left ventricular remodeling disparities between genders | baseline; 3 months and 1 year after myocardial infarction onset
  The primary outcome measure will be the occurrence of left ventricular remodeling (defined as a change in ventricular volume of more than 10% during follow-up) measured with cardiac imaging (echocardiography and MRI)

SECONDARY OUTCOMES:
Evaluate the evolution of remodeling at Month 3 | 3 months
  Changes in ventricular volumes between acute phase and 3 months measured with cardiac imaging (echocardiography and MRI)
Assess remodeling changes between inclusion and Month 12 | 1 year
  Changes in ventricular volumes between acute phase and 1 year measured with cardiac imaging (echocardiography and MRI)
Assess the prevalence of comorbidities and their impact on the effect on the outcome: post-infarction cardiac remodeling with gender (cardiovascular risk factors, renal function, hepatic functionperipheral artery disease, way of life) | 3 months and 1 year
  renal function: uremia and creatinine levels, combined with an assessment of the protein-to-creatinine ratio in urine samples, and a cyto-bacteriological examination of urine to detect hematuria; hepatic function: The Fibroscan® is a device that enables a non-invasive and efficient assessment of liver fibrosis and steatosis within minutes at the patient's bedside, providing an immediate result displayed on the device screen; peripheral artery disease: Doppler echocardiography of the supra-aortic trunks; way of life : dietetary, stress and physical activity scores common CV risk factors: prior history of hypertension, hypercholesterolaemia, tobacco use, diabetes
Explore prognostic disparities between men and women. | yearly, up to 10 years
  Occurrence of complications and cardiovascular events (cardiovascular death, heart failure, stroke, or reinfarction)
Evaluate lifestyle habits up to 10 years: outcome anxiety/depression | yearly, up to 10 years
  Anxiety/Depression (A.D) score: 2 scales from 0 to 21, the greatest the more prone to either anxiety or depression
Evaluate lifestyle habits up to 10 years: outcome diet score | yearly, up to 10 years
  Mediteranean diet score (MED): from 0 to 14, the greatest the more relevant for mediteranean diet
Evaluate lifestyle habits up to 10 years: outcome physical activity | yearly, up to 10 years
  physical activity: lipid research clinics (LRC); 2 scales from 1 to 5, the greatest the less active
Assess the risk of remodeling based on specific parameters in female subjects: presence of endometriosis | baseline
  presence or absence of endometriosis
Assess the risk of remodeling based on specific parameters in female subjects: presence of polycystic ovary | baseline
  presence or absence of polycystic ovary
Assess the risk of remodeling based on specific parameters in female subjects: presence of uterine fibroma | baseline
  presence or absence of uterine fibroma
Assess the risk of remodeling based on specific parameters in female subjects: presence of hormonal therapy | baseline
  presence or absence of hormonal therapy
Assess the risk of remodeling based on specific parameters in female subjects: date of first period | baseline
  date of first period
Assess the risk of remodeling based on specific parameters in female subjects: pregnancy | baseline
  number of pregnancy
Assess the risk of remodeling based on specific parameters in female subjects: children | baseline
  number of children
Assess the risk of remodeling based on specific parameters in female subjects: obstetrical event | baseline
  absence or presence of obstetrical events (hypertension, diabete, microsomia and macrosomia)
Assess the risk of remodeling based on specific parameters in female subjects: menopause | baseline
  absence or presence of menopause

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Angers, Angers, France